CLINICAL TRIAL: NCT01101152
Title: Effectiveness of the Dual Serotonin Norepinephrine Reuptake Inhibitor Desvenlafaxine Succinate in Healthy Females and Males
Brief Title: Effectiveness of the Dual Serotonin Norepinephrine Reuptake Inhibitor Desvenlafaxine Succinate in Healthy Volunteers
Acronym: DVS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Pierre Blier, MD, Ph.D., University of Ottawa Institute of Mental Health Research
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: REB-2009036
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: Antidepressant; healthy volunteers; desvenlafaxine succinate; norepinephrine reuptake; serotonin reuptake; tyramine test
MeSH Terms: interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Female (Experimental)
  Interventions: Drug: Desvenlafaxine succinate
- Male (Experimental)
  Interventions: Drug: Desvenlafaxine succinate

INTERVENTIONS:
Drug: Desvenlafaxine succinate — Tablets of 50 mg,100 mg; Dosing regimen: 50, 100, 200 mg/day; 1 week for each dose regimen;
  1 tablet a day for doses of 50 and 100mg/day, and 2 tablets of 100mg for dose of 200mg/day
  Other Names: Pristiq

SUMMARY:
DVS is the main metabolite of the antidepressant/anxiolytic medication Venlafaxine (Effexor). Like parent compound, DVS is an antidepressant inhibiting both serotonin (5-HT) and norepinephrine (NE) reuptake. However, no studies to date describe the in vivo potency of this drug on monoamines reuptake. Consequently, it appears essential to determine the potency of DVS in human subjects using a wide dose range in order to determine at which dose(s) it starts inhibiting 5-HT and NE reuptake. The investigators are interested in learning whether there is a gender difference in the dose of the study medication at which NE reuptake inhibition occurs.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects between 18 and 40 years of age, including those on oral contraceptive pills
* Male subjects between 18-40 years of age
* Written informed consent signed by the subject.

Exclusion Criteria:

* Life-time personal history of diagnosis of major depression according to the DSM-IV (American Psychiatry Association, 1994) using the MINI (Sheehan et al. 1998)
* Blood pressure greater than 140/90 and a pulse rate greater than 90bpm
* Evidence of significant physical illness contraindicating the use of DVS, found on physical or in the laboratory data obtained during the first week of the study
* Obvious mental retardation rendering the response to investigators unreliable
* Pregnancy, or absence of adequate contraceptive method.
* Concurrent use of psychotropic medication such as antipsychotics, mood stabilizers or regular use of benzodiazepines.
* Participation in a clinical trial within 30 days of entry into the current study
* Intolerance to Desvenlafaxine

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The degree of norepinephrine reuptake in response to the increasing levels of the study medication will be assessed and compared between genders | 1 month

SECONDARY OUTCOMES:
The degree of serotonin reuptake in response to the increasing levels of the study medication will be assessed and compared between genders | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Blier, M.D., Ph.D., Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa Institute of Mental Health Research, Ottawa, Ontario, Canada

REFERENCES:
- See also: University of Ottawa Institute of Mental Health Research homepage — http://www.imhr.ca